CLINICAL TRIAL: NCT05770765
Title: Creation of a Bank of Biological Materials and Associated Data Related to Patients With Infectious and Tropical Diseases
Acronym: TropicaBiobank
Status: Recruiting | Type: Observational
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-46
Record Dates: First submitted 2023-03-02; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 40 Years
Biospecimen Retention: Samples With DNA — The type of samples collected and stored in the biobank consists of human biological matrices liquids and solids, DNA, protein extracts or subcellular fractions, bacterial isolates and arthropods taken from patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is the protocol that formalizes the establishment of the TROPICA-BIOBANK biobank

DETAILED DESCRIPTION:
Subjects who will access the Department of Infectious and Tropical Diseases for investigations, analyzes or visits on suspicion of infectious or tropical disease, hospitalized patients and/or patients participating in proposed clinical trials from the Department will be enrolled. Healthy volunteer donors may also be enrolled.

The type of samples collected and stored in the biobank consists of human biological matrices liquids and solids, DNA, protein extracts or subcellular fractions, bacterial isolates and arthropods taken from patients. The collection of samples takes place through the support of various professional figures (doctor, nurse, laboratory technician, biologist/biotechnologist) together with associated data.

The samples are de-identified and protected by an encryption system (through the system computer diagnostic data management of the laboratory of the IRCCS Sacro Cuore Don Calabria) and stored at a temperature of -80°C, in the Department's freezers. Samples are stored for 40 years. In order to monitor the quality of the samples over the storage time, a selection of samples used as monthly analytical quality controls will be retested periodically (every 10 years). At the end of the storage time, it will be evaluated whether to extend the storage time of the unused biological samples and associated data or if these will be destroyed. In the first case, an amendment to this Protocol will be submitted to the CESC for approval, in which will specify the duration of the extension of the conservation of the samples and associated data. In the second case, no further data will be collected on the aforementioned samples, without prejudice to their use of those possibly already collected to determine, without altering them, the results of searches already in progress.

The samples will in any case be destroyed if they are not in good condition.

ELIGIBILITY:
Inclusion Criteria:

• Informed consent (for healthy volounteers also: age > 18 years, health status ascertained by laboratory tests, electrocardiogram and medical examination)

Exclusion Criteria:

* History of alcohol/drug abuse
* Pregnant or breastfeeding women, unless there are justified and documented needs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who access the Department for investigations, analyzes or visits on suspicion infectious or tropical disease, hospitalized patients and/or patients participating in proposed clinical trials from the Department will be enrolled . Healthy volunteer donors may also be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2059-10-30 (Estimated); Study Completion 2059-10-30 (Estimated)

PRIMARY OUTCOMES:
Presence of a viral, bacterial or parasitic pathogen | 40 years
  Result of laboratory tests on the pathogen responsible for the disease of interest

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Sacro Cuore Don Calabria hospital, Negrar, Verona, Italy